CLINICAL TRIAL: NCT04264052
Title: The Feasibility of Continuous Bronchoscopy During Exercise in Healthy Adults in Assessing Large Airways Collapse
Brief Title: Characterisation of Large Airway Collapse During Exercise (LACE)
Acronym: LACE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Imperial College London (Other)
Collaborators: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 19IC5362
Record Dates: First submitted 2019-09-19; First posted 2020-02-11 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Airway Disease
Keywords: excessive dynamic airway collapse; tracheobronchomalacia; large airways collapse
MeSH Terms: conditions — Tracheobronchomalacia | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CBE & MRI: Forty healthy volunteers split in different age ranges (20-30 years n=10, 30-40 years n=10, 40-50 years n=10 and 50-60 years n=10) will undergo two airway assessments at rest and during exercise. The exercise assessments will be a continuous bronchoscopy during exercise (CBE-1st visit) and magnetic resonance imaging (MRI-2nd visit) separated by at least three days to ensure for a sufficient cardiorespiratory and musculoskeletal recovery.
  Interventions: Diagnostic Test: CBE & MRI

INTERVENTIONS:
Diagnostic Test: CBE & MRI — The diagnostic tests will be consisted by two visits.
  In the first visit participants will undergo a medical history assessment and they will complete questionnaires related to the lung function (MRC Dyspnoea score, Dyspnoea-12 questionnaire, and Visual Analogue Scale). A spirometry will be performed to assess the lung function. Bronchoscopy will be performed at rest in a semi-supine position (on a reclined bed) and then during exercise on a treadmill.
  In the second visit, spirometry and questionnaires will be performed prior to resting and during exercise measurements on a magnetic resonance imaging (MRI) scan.
  Rest: Structural imaging of the neck and chest will be performed followed by dynamic imaging of the airways during several inspiratory and expiratory manoeuvres. No IV contrast media will be used.

SUMMARY:
The large central airways (i.e. trachea and bronchi) act as a conduit to enable lower airway ventilation but also facilitate airway clearance during dynamic manoeuvres, such as coughing. It is becoming increasingly well recognised however, that in a significant proportion of individuals with chronic airway disease (e.g. chronic obstructive pulmonary disease-COPD or chronic asthma) and in those with an elevated body mass index (BMI), that the large airways may exhibit a tendency to excessive closure or narrowing. This large airway collapse (LAC) can be associated with exertional breathlessness and difficulty clearing airway secretions. A variety of terms have been used to describe LAC including excessive dynamic airway collapse (EDAC) or if the cartilaginous structures are involved then tracheobronchomalacia (TBM).

One clear limitation of the current approach to diagnosis is the fact that many of the 'diagnostic' tests employed, utilise static, supine measures +/- forced manoeuvres. These are somewhat physiologically flawed and differ markedly from the reality of the heightened state of airflow that develops during exertion. i.e. forced manoeuvres likely induce very different turbulent and thoracic pressure changes, in contrast to the hyperpnoea of real-life physical activity (i.e. walking or cycling). A current unanswered question is therefore, what happens to the large airway dynamic movement of healthy individuals (and ultimately patients) during real-life exercise and how does this compare with the measures taken during a forced manoeuvre, either during a bronchoscopy or during an imaging study such as CT or MRI scan.

The key aim of this study is therefore to evaluate and characterise large airway movement in a cohort of healthy adults during a real-life exercise challenge and to compare this with findings from a dynamic expiratory MRI. In order to achieve this, the investigators proposes to develop and test the feasibility of an exercise-bronchoscopy protocol.

DETAILED DESCRIPTION:
The large central airways (i.e. trachea and bronchi) act as a conduit to enable lower airway ventilation but also facilitate airway clearance during dynamic manoeuvres, such as coughing. It is becoming increasingly well recognised however, that in a significant proportion of individuals with chronic airway disease (e.g. chronic obstructive pulmonary disease or chronic asthma) and in those with an elevated body mass index (BMI), that the large airways may exhibit a tendency to excessive closure or narrowing. This large airway collapse (LAC) can be associated with exertional breathlessness and difficulty clearing airway secretions. A variety of terms have been used to describe LAC including excessive dynamic airway collapse (EDAC) or if the cartilaginous structures are involved then tracheobronchomalacia (TBM).

At the current time, there is considerable debate regarding the definition of LAC. Typically the 'excessive' collapse underpinning a 'diagnosis' of EDAC is defined as excessive bulging of the posterior tracheal membrane into the airway lumen during expiration without associated collapse of the cartilaginous rings, however the degree to which the trachea closes, to constitute EDAC is debated, with literature varying from >50% to >90%. Moreover, partial expiratory airways collapse (up to 50% reduction in airways cross-sectional area) can be identified in 70-80% of healthy individuals during dynamic computed tomography (CT).

One clear limitation of the current approach to diagnosis is the fact that many of the 'diagnostic' tests employed, utilise static, supine measures +/- forced manoeuvres. These are somewhat physiologically flawed and differ markedly from the reality of the heightened state of airflow that develops during exertion. i.e. forced manoeuvres likely induce very different turbulent and thoracic pressure changes, in contrast to the hyperpnoea of real-life physical activity (i.e. walking or cycling). A current unanswered question is therefore, what happens to the large airway dynamic movement of healthy individuals (and ultimately patients) during real-life exercise and how does this compare with the measures taken during a forced manoeuvre, either during a bronchoscopy or during an imaging study such as CT or MRI scan.

The key aim of this study is therefore to evaluate and characterize large airway movement in a cohort of healthy adults during a real-life exercise challenge and to compare this with findings from a dynamic expiratory MRI and MRI during exercise. In order to achieve this, the investigators propose to develop and test the feasibility of an exercise-bronchoscopy protocol.

As a clinical service, the investigators have extensive experience of evaluating movement of the upper airway and larynx during strenuous exercise. The Principal Investigator currently performs over 100 continuous laryngoscopy during exercise (CLE) tests per year, whereby a small laryngoscope is placed in the upper airway and is secured on a headgear to allow visualisation of the laryngeal and subglottic movement during exercise. i.e. whilst a subject performs running exercise. This test has an established role in patient evaluation and a proven safety record in the assessment of laryngeal closure during exercise. The research team has performed approximately 500 CLE tests in the Royal Brompton Hospital, with no serious adverse outcome.

The investigators thus now propose to utilise a similar exercise technique but to advance the scope (using a bronchoscope because this is needed to evaluate the lower airways) slightly more distally to allow visualisation of the large airways during an exercise challenge. Others have also utilised a similar approach. Specifically, a study evaluated military personal with symptoms of exertional dyspnoea. As part of this study the research team performed dynamic bronchoscopy with real-time observation on a bicycle ergometer.

Therefore, the investigators recommend the application of a similar approach, termed continuous bronchoscopy during exercise (CBE) to evaluate large airway movement during exercise and to report the feasibility and tolerability of the technique and to compare findings with imaging techniques (i.e. as is often used to diagnose EDAC) using MRI. In this initial study however, the investigators propose to study only healthy subjects to assess feasibility and provide comparator data for later work. i.e. to use this data to provide pilot feasibility work and thus to utilise results to inform and power later work, as indicated.

Study Rationale The investigators hypothesise that exercise bronchoscopy is feasible to perform for the investigation of EDAC. It is also hypothesised that findings on dynamic static manoeuvres (i.e. when subjects are asked to perform a forced dynamic breath out) with both a bronchoscope in situ and also during MRI will exaggerate a tendency to closure and not relate to the real-life physiological airway stress encountered during exercise.

STUDY OBJECTIVES

The primary objective of this study is to investigate the feasibility and safety of continuous bronchoscopy during exercise.

The following hypothesis will be tested:

1. Continuous bronchoscopy during exercise is feasible
2. Continuous bronchoscopy during exercise is well-tolerated
3. Continuous bronchoscopy during exercise provides stable large airway images; to enable reliable assessment of any propensity to large airway collapse.

Secondary objectives include:

1. To evaluate the degree of LAC apparent in normal subjects during exercise and to compare this with static forced expiratory manoeuvres in MRI.
2. To evaluate the degree of LAC from MRI in normal subjects during forced expiratory manoeuvres.

To compare findings between modalities and to compare all findings with simple baseline physiological measures, such as lung function.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will need to be within the age range of 20-60 years old
* have no known respiratory disease and normal spirometry
* be able to exercise without medical reason for limitation.

Exclusion Criteria:

* Subjects who have a significant comorbidity that prohibit exercise
* have had a respiratory infection within the last month
* known respiratory disease
* current smokers or are pregnant.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects will be healthy and ≥ 20 to 60 years old.
  The total sample size will be 40 subjects. 10 for each age group (20-30; 30-40; 40-50; 50-60 years).
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Feasibility of continuous bronchoscopy during exercise (CBE): questionnaire | 12 months
  Primary outcome will be the feasibility of continuous bronchoscopy during continuous exercise in healthy adults. Feasibility will be assessed via a post CBE tolerability questionnaire.
  The post exercise tolerability questionnaire aims to evaluate the upper airways function during exercise and the discomfort that the participant might experience during the test. It consists of 5 questions (Part A) where the score ranges from 1 (strongly disagree) to 5 (strongly agree), and 2 questions (Part B) where the score ranges from 1 (None at all) to 10 (Unbearable amount).
  The total score that will confirm the feasibility of CBE should be < 3 or < 5, for Part A and B, respectively.
  The questions relate to the tolerability of the CBE test (e.g., Exercise with the camera in place cause discomfort, 1 (strongly agree) to 5 (strongly disagree).

SECONDARY OUTCOMES:
Diagnostic capacity of CBE and MRIE | 12 months
  To evaluate the degree of large airway collapse (LAC) apparent in normal subjects via continuous bronchoscopy during exercise (CBE) and to compare this with static forced expiratory manoeuvres in magnetic resonance imaging (MRI) and MRI during exercise (MRIE).
  Flexible bronchoscopy and MRI at rest will be performed using dynamic inspiratory and expiratory manoeuvres.
  CBE will be performed on a treadmill utilising a linear individualised ramp protocol. Heart rate and electrocardiogram will be monitored throughout the test.
  The degree of LAC will be estimated in percentage reduction of the airway lumen in several sites of the trachea and main bronchi. In bronchoscopy the reduction will be classified as 0 to 50% / 50 to 75% / 75 to 100% / 100% airway closure. In MRI LAC will be diagnosed as >50% airway closure.
Comparing dynamic versus physical exertion large airway collapse in CBE and MRIE | 12 months
  To estimate the percentage of LAC from MRI in normal subjects during forced expiratory manoeuvres at rest and during exercise for both modalities.
  More specifically, the reduction (%) of LAC will be estimated in bronchoscopy at rest and will be compared with CBE to evaluate whether physical exertion can induce the similar response to dynamic expiratory manoeuvres. Similarly, percentage of LAC will be estimated in MRI at rest.
  Comparisons will be performed using statistical tests (e.g., Paired sample T-tests).
Exploring the diagnostic capacity of different exercise modalities to assess LAC | 12 months
  To compare findings between modalities (treadmill vs dynamic MRI images.
  The percentages of LAC between CBE and MRI will be compared (via statistical tests such as t-tests and Pearson's correlation tests.

CONTACTS AND LOCATIONS:
Overall Officials: James Hull, Dr, Principal Investigator — Royal Brompton Hospital-Imperial College London
Locations (1):
- Royal Brompton Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No